CLINICAL TRIAL: NCT02535195
Title: Effect of Ginger Supplement on Non-alcoholic Fatty Liver
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr Azita Hekmatdoost (Other)
Responsible Party: Sponsor-Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93-03-161-27265
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ginger (Active Comparator): Participants were randomly divided based on age, sex and severity of steatosis in two groups. Randomization lists were computer-generated by a statistician and participants, project managers and employees at the clinic were completely unaware (blind) about intervention and control groups. At the first visit, baseline data were gathered and patients advised to consume 2 capsules content 500 mg of ginger (made in Green Plants of Life Pharmaceutics Co., Iran) or placebo (starch) one hour after breakfast and two capsules after dinner for 3 weeks. Capsules was administrated for all patients in the first week for 3 weeks and in each visit new series of supplement was prescribed.
  Interventions: Dietary Supplement: Ginger supplement
- Placebo (Placebo Comparator): 2 capsules content 500 mg of placebo(starch) (made in Green Plants of Life Pharmaceutics Co., Iran) one hour after breakfast and two capsules after dinner for 3 weeks. Capsules was administrated for all patients in the first week for 3 weeks and in each visit new series of supplement was prescribed.
  Interventions: Dietary Supplement: Placebo (starch)

INTERVENTIONS:
Dietary Supplement: Ginger supplement
  Arms: Ginger
Dietary Supplement: Placebo (starch)
  Arms: Placebo

SUMMARY:
The hypothesis of this study was that ginger supplement consumption can be introduced as a new therapeutic strategy for non-alcoholic fatty liver disease through the improved body antioxidant activity, reduced levels of inflammation and insulin resistance. A randomized double-blind study was designed to evaluate this hypothesis in order to examine the effectiveness of ginger supplement in patients with non-alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* presence of steatosis on ultrasound examination
* high concentration of liver enzyme (alanine aminotransferase (ALT) greater than normal range of 1.5 times)

Exclusion Criteria:

* various types of hepatitis
* diabetes mellitus
* cancer inherited disorders affecting liver condition (storage disorders of iron, copper, and others)
* non-treated hypothyroidism
* using alcohol
* consumption of phenytoin amoxyfan and lithium
* using minerals multivitamin supplements such as vitamin E, vitamin D, supplements made from Silybum marianum extract like livergol
* weight loss surgery in the last year or strict diets to weight loss in the past three months pregnancy
* lactation
* autoimmune diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Serum levels of the ALT liver enzyme | 12 weeks
Serum levels of the AST liver enzyme | 12 weeks

SECONDARY OUTCOMES:
controlled attenuation parameter(CAP) score | 12 weeks
  controlled attenuation parameter(CAP) score is a novel measurement for evaluation of hepatic steatosis and it evaluated in dB/m at 3.5 MHz by M probe. normal range is 100- 140 dB/M.